CLINICAL TRIAL: NCT02531438
Title: A Phase 3 Randomized, Double-Blind, Multi-Center Study to Compare the Safety and Efficacy of Omadacycline Intravenous (IV)/Oral (PO) to Moxifloxacin IV/PO for Treating Adults Subjects With Community-Acquired Bacterial Pneumonia
Brief Title: Omadacycline vs Moxifloxacin for the Treatment of CABP (EudraCT #2013-004071-13)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-CABP-1200
Record Dates: First submitted 2015-07-14; First posted 2015-08-24 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Bacterial Pneumonia; Community-Acquired Infections
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Infections | interventions — omadacycline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omadacycline (Experimental): Omadacycline IV; Omadacycline tablets
  Interventions: Drug: Omadacycline
- Moxifloxacin (Active Comparator): Moxifloxacin IV; Moxifloxacin tablets
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Omadacycline — Injection for IV; Oral tablets
  Arms: Omadacycline
Drug: Moxifloxacin — IV solution; Oral tablets
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of omadacycline as compared to moxifloxacin in the treatment of adults with community-acquired bacterial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ages 18 years or older who have signed the informed consent
* Has qualifying bacterial pneumonia
* Female patients must not be pregnant at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Known or suspected hospital-acquired pneumonia
* Evidence of significant immunological disease
* Has a history of hypersensitivity or allergic reaction to any tetracycline or to any fluoroquinolone antibiotic
* Has received an investigational drug within past 30 days
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-02-05 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (140):
- United States (12):
  - Site 514, Birmingham, Alabama
  - Site 501, Mobile, Alabama
  - Site 508, Laguna Hills, California
  - Site 505, Ventura, California
  - Site 513, Stamford, Connecticut
  - Site 511, Zachary, Louisiana
  - Site 503, Detroit, Michigan
  - Site 520, Saint Paul, Minnesota
  - Site 512, St Louis, Missouri
  - Site 506, Buffalo, New York
  - Site 509, Dayton, Ohio
  - Site 516, Huntington, West Virginia
- Site 220, Liège, Belgium
- Brazil (4):
  - Site 276, Belo Horizonte, Minas Gerais
  - Site 277, Passo Fundo, Rio Grande do Sul
  - Site 274, Porto Alegre, Rio Grande do Sul
  - Site 279, São José do Rio Preto, São Paulo
- Bulgaria (7):
  - Site 305, Kyustendil
  - Site 303, Pernik
  - Site 304, Plovdiv
  - Site 306, Sliven
  - Site 301, Sofia
  - Site 302, Sofia
  - Site 307, Sofia
- Croatia (8):
  - Site 250, Požega
  - Site 205, Slavonski Brod
  - Site 212, Zadar
  - Site 201, Zagreb
  - Site 202, Zagreb
  - Site 203, Zagreb
  - Site 251, Zagreb
  - Site 405, Zagreb
- Czechia (4):
  - Site 412, Kyjov
  - Site 410, Prague
  - Site 411, Prague
  - Site 414, Třebíč
- Georgia (5):
  - Site 390, Tbilisi
  - Site 391, Tbilisi
  - Site 392, Tbilisi
  - Site 393, Tbilisi
  - Site 394, Tbilisi
- Germany (3):
  - Site 415, Heidelberg
  - Site 416, Jena
  - Site 417, Paderborn
- Greece (5):
  - Site 207, Athens, Attica
  - Site 420, Athens, Attica
  - Site 210, Athens
  - Site 421, Athens
  - Site 208, Thessaloniki
- Hungary (7):
  - Site 310, Budapest
  - Site 311, Budapest
  - Site 312, Budapest
  - Site 314, Debrecen
  - Site 316, Miskolc
  - Site 313, Nyíregyháza
  - Site 315, Székesfehérvár
- Israel (5):
  - Site 213, Holon
  - Site 214, Nazareth
  - Site 217, Petah Tikva
  - Site 215, Ramat Gan
  - Site 216, Safed
- Latvia (4):
  - Site 322, Daugavpils
  - Site 323, Liepāja
  - Site 320, Riga
  - Site 321, Riga
- Mexico (5):
  - Site 228, Guadalajara, Jalisco
  - Site 472, Guadalajara, Jalisco
  - Site 227, Monterrey, Nuevo León
  - Site 471, Monterrey, Nuevo León
  - Site 230, Xalapa, Veracruz
- Peru (7):
  - Site 234, Cusco
  - Site 233, Lima
  - Site 236, Lima
  - Site 238, Lima
  - Site 239, Lima
  - Site 481, Lima
  - Site 237, Trujillo
- Philippines (5):
  - Site 555, Caloocan
  - 552, Iloilo City
  - 554, Manila
  - Site 551, Quezon City
  - Site 553, Quezon City
- Poland (5):
  - Site 332, Chrzanów
  - Site 333, Katowice
  - Site 330, Lodz
  - Site 331, Wroclaw
  - Site 334, Łęczna
- Romania (6):
  - Site 344, Brasov
  - Site 340, Bucharest
  - Site 342, Bucharest
  - Site 343, Bucharest
  - Site 345, Craiova
  - Site 341, Timișoara
- Russia (10):
  - 352, Moscow
  - Site 350, Moscow
  - Site 351, Moscow
  - Site 353, Saint Petersburg
  - Site 354, Saint Petersburg
  - Site 355, Saint Petersburg
  - Site 356, Saint Petersburg
  - 357, Sestroretsk
  - Site 358, Vsevolozhsk
  - Site 359, Zelenograd
- Slovakia (4):
  - Site 431, Bratislava
  - Site 430, Levice
  - Site 432, Martin
  - Site 433, Nitra
- South Africa (6):
  - Site 241, Benoni, Gauteng
  - Site 436, Centurion, Gauteng
  - Site 242, Pretoria, Guateng
  - Site 244, Thabazimbi, Limpopo
  - Site 245, Middelburg, Mpumalanga
  - Site 437, Somerset West, Western Cape
- South Korea (4):
  - Site 293, Daegu
  - Site 291, Seoul
  - Site 292, Seoul
  - Site 294, Seoul
- Spain (5):
  - Site 225, Elche, Alicante
  - Site 221, Barcelona, Catalonia
  - Site 440, Barcelona, Catalonia
  - Site 224, Alzira, Valencia
  - Site 226, Alicante
- Taiwan (5):
  - Site 299, Kaohsiung City
  - Site 297, Tainan
  - Site 295, Taipei
  - Site 296, Taipei
  - Site 298, Taipei
- Turkey (Türkiye) (4):
  - Site 247, Ankara
  - Site 248, Ankara
  - Site 249, Ankara
  - Site 246, Trabzon
- Ukraine (9):
  - Site 380, Dnipro
  - Site 373, Dnipropetrovsk
  - Site 374, Kharkiv
  - Site 375, Kharkiv
  - Site 370, Kyiv
  - Site 372, Kyiv
  - Site 378, Kyiv
  - Site 379, Kyiv
  - Site 376, Zaporizhia

REFERENCES:
- [Derived] Rodriguez GD, Warren N, Yashayev R, Chitra S, Amodio-Groton M, Wright K. Omadacycline in the treatment of community-acquired bacterial pneumonia in patients with comorbidities: a post-hoc analysis of the phase 3 OPTIC trial. Front Med (Lausanne). 2023 Jul 28;10:1225710. doi: 10.3389/fmed.2023.1225710. eCollection 2023. PMID 37575994
- [Derived] Vacalis S, Brunton S, Gindi J. Omadacycline in Skin Infections and Pneumonia: A Review of the Evidence. J Fam Pract. 2022 Jun;71(5 Suppl):S10-S21. doi: 10.12788/jfp.0424. PMID 35776862
- [Derived] Cornely OA, File TM Jr, Garrity-Ryan L, Chitra S, Noble R, McGovern PC. Safety and efficacy of omadacycline for treatment of community-acquired bacterial pneumonia and acute bacterial skin and skin structure infections in patients with mild-to-moderate renal impairment. Int J Antimicrob Agents. 2021 Feb;57(2):106263. doi: 10.1016/j.ijantimicag.2020.106263. Epub 2020 Dec 14. PMID 33326848
- [Derived] Ramirez JA, Tzanis E, Curran M, Noble R, Chitra S, Manley A, Kirsch C, McGovern PC. Early Clinical Response in Community-acquired Bacterial Pneumonia: From Clinical Endpoint to Clinical Practice. Clin Infect Dis. 2019 Aug 1;69(Suppl 1):S33-S39. doi: 10.1093/cid/ciz397. PMID 31367741
- [Derived] Stets R, Popescu M, Gonong JR, Mitha I, Nseir W, Madej A, Kirsch C, Das AF, Garrity-Ryan L, Steenbergen JN, Manley A, Eckburg PB, Tzanis E, McGovern PC, Loh E. Omadacycline for Community-Acquired Bacterial Pneumonia. N Engl J Med. 2019 Feb 7;380(6):517-527. doi: 10.1056/NEJMoa1800201. PMID 30726692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant randomization was stratified by Pneumonia Outcomes Research Team (PORT) Risk Class (II or III/IV), receipt of an allowed antibacterial therapy in the 72 hours prior to study treatment, and geographic region. All participants were expected to present with CABP severe enough to require at least 3 days of intravenous (IV) treatment.
Pre-assignment Details: Participants who met inclusion criteria and did not meet exclusion criteria were randomly assigned to a treatment group, and received their first dose of test article within 4 hours after randomization. All participants were expected to present with CABP PORT Risk Class II, III, or IV to require a minimum of at least 3 days of IV treatment.
Groups:
- Omadacycline: Participants received omadacycline 100 milligrams (mg) intravenously (IV) every 12 hours (q12h) (first 2 doses), followed by 100 mg IV every 24 hours (q24h) (starting 24 hours after the first dose), with the option to switch to a 300 mg (two 150 mg omadacycline tablets and 1 over-encapsulated placebo tablet matching moxifloxacin) oral administration q24h after at least 3 days (4 doses) of IV treatment. The total duration of test article therapy (IV plus oral administration) for all participants was at least 7 days and no more than 14 days.
- Moxifloxacin: Participants received moxifloxacin 400 mg IV q24h (with a single placebo infusion to match the omadacycline dosing regimen 12 hours after the first dose on Day 1) with the option to switch to a 400 mg (one 400 mg moxifloxacin over-encapsulated tablet and 2 placebo tablets matching omadacycline tablets) oral administration q24h after at least 3 days (4 doses) of IV treatment. The total duration of test article therapy (IV plus oral administration) for all participants was at least 7 days and no more than 14 days.
Period: Overall Study
Arm/Group | Omadacycline | Moxifloxacin
Started | 386 | 388
Completed | 356 | 362
Not Completed | 30 | 26
Not completed — Adverse Event | 7 | 9
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Death | 6 | 3
Not completed — Randomized, but Not Treated | 4 | 0
Not completed — Missed EOT/PTE Visit | 5 | 2
Not completed — Randomized with Exclusion Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline | Moxifloxacin | Total
Number analyzed (Participants) | 386 | 388 | 774
Age, Customized [Count of Participants; unit: Participants]
  18 to 45 years old | 62 | 61 | 123
  >45 to 65 years old | 172 | 155 | 327
  >65 years old | 152 | 172 | 324
  >75 years old | 75 | 83 | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 169 | 347
  Male | 208 | 219 | 427
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 17 | 18 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 7 | 18
  White | 356 | 355 | 711
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Clinical Response
Description: Early clinical response is defined as clinical success, categorized by survival with improvement of at least 1 level compared to Baseline in at least 2 CABP symptoms (cough, sputum production, pleuritic chest pain, and dyspnea) with no worsening in the other CABP symptoms. Response was determined programmatically using the investigator's assessment of the CABP symptoms. The severity of the participant's CABP symptoms was evaluated on a 4-point scale (absent, mild, moderate, or severe) based upon the CABP Subject Symptom Severity Guidance Framework for Investigator Assessment. An indeterminate response is defined as one that could not be adequately inferred because the participant was not assessed because they withdrew consent, were lost to follow-up, or other specified reason. Clinical failure is defined as no improvement by at least 1 level in CABP symptoms, worsening of any CABP symptom, alternative antibacterial treatment for CABP, discontinuation due to adverse event, or death.
Time Frame: Screening; 72 to 120 hours after the first dose of test article
Population: Intent-to-Treat (ITT) Population: all randomized participants regardless of whether or not the participant received the test article
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Moxifloxacin
Number analyzed (Participants) | 386 | 388
Participants
  Clinical success | 313 | 321
  Clinical failure | 49 | 47
  Indeterminate | 24 | 20
Statistical Analysis 1: Comparison: Omadacycline vs Moxifloxacin; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = -1.6, 95% CI 2-sided [-7.1 to 3.8] — The 95% confidence interval was constructed based on the Miettinen and Nurminen method without stratification. Treatment difference for a response of clinical success was calculated as omadacycline minus moxifloxacin

2. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Clinical Response in the ITT Population at the Post Therapy Evaluation (PTE) Visit
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: survival after completion of a test article regimen without receiving any systemic antibacterial therapy other than test article, resolution of signs/symptoms of the infection present at Screening with no new symptoms/complications attributable to CABP and no need for further antibacterial therapy. Clinical Failure: alternative antibacterial treatment for CABP was required prior to the PTE Visit related to either (a) progression/development of new CABP symptoms or (b) development of infectious complications of CABP. Other reasons for clinical failure: participant received antibiotics that may have been effective for the infection under study for a different infection from the one under study; death prior to the PTE Visit. Indeterminate: the clinical response to test article could not be adequately inferred.
Time Frame: Screening; 5 to 10 days after the last day of therapy
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Moxifloxacin
Number analyzed (Participants) | 386 | 388
Participants
  Clinical success | 338 | 330
  Clinical failure | 32 | 42
  Indeterminate | 16 | 16
Statistical Analysis 1: Comparison: Omadacycline vs Moxifloxacin; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 2.5, 95% CI 2-sided [-2.4 to 7.4] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Clinical Response in the Clinically Evaluable-Post Therapy Evaluation (CT-PTE) Population
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: survival after completion of a test article regimen without receiving any systemic antibacterial therapy other than test article, resolution of signs/symptoms of the infection present at Screening with no new symptoms/complications attributable to CABP and no need for further antibacterial therapy. Clinical Failure: alternative antibacterial treatment for CABP was required prior to the PTE Visit related to either (a) progression/development of new CABP symptoms or (b) development of infectious complications of CABP. Other reasons for clinical failure: participant received antibiotics that may have been effective for the infection under study for a different infection from the one under study; death prior to the PTE Visit.
Time Frame: Screening; 5 to 10 days after the last day of therapy
Population: CE-PTE Population: all participants in the ITT Population meeting additional pre-defined criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Moxifloxacin
Number analyzed (Participants) | 340 | 345
Participants
  Clinical success | 316 | 312
  Clinical failure | 24 | 33
Statistical Analysis 1: Comparison: Omadacycline vs Moxifloxacin; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 2.5, 95% CI 2-sided [-1.7 to 6.8] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the signing of Informed Consent Form to the time of the Final Follow-up assessment (up to 30 to 37 days after the start of the first infusion of test article)
Description: Adverse events are reported for members of the Safety Population, comprised of all randomized participants who received test article (either active or placebo). Treatment-emergent adverse events, defined as events occurring after the first dose of active test article, are reported.
Arm/Group | Omadacycline | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 8/382 | 4/388
Serious Adverse Events (participants affected / at risk) | 23/382 | 26/388
Other Adverse Events (participants affected / at risk) | 63/382 | 94/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=382) | Moxifloxacin (N=388)
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Cardiogenic Shock (Cardiac disorders) | 2 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatic Congestion (Hepatobiliary disorders) | 0 | 1
Influenza (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 2 | 6
Cellulitis (Infections and infestations) | 1 | 0
Infectious Pleural Effusion (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 1 | 2
Atypical Mycobacterial Pneumonia (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 2
human Immunodeficiency Virus (HIV) Infection (Infections and infestations) | 0 | 1
Infective Exacerbation Of Bronchiectasis (Infections and infestations) | 0 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 1
Bladder Injury (Injury, poisoning and procedural complications) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic Aneurysm Rupture (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=382) | Moxifloxacin (N=388)
Vomiting (Gastrointestinal disorders) | 10 | 6
Constipation (Gastrointestinal disorders) | 9 | 6
Nausea (Gastrointestinal disorders) | 9 | 21
Diarrhea (Gastrointestinal disorders) | 4 | 31
Alanine aminotransferase increased (Investigations) | 14 | 18
Gamma-glutamyl transferase increased (Investigations) | 10 | 8
Aspartate aminotransferase increased (Investigations) | 8 | 14
Headache (Nervous system disorders) | 8 | 5
Insomnia (Psychiatric disorders) | 10 | 8
Hypertension (Vascular disorders) | 13 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication and require the removal of confidential information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT02531438/Prot_SAP_000.pdf